CLINICAL TRIAL: NCT00849524
Title: A Phase II Study of Repeat Intranodal Injections of Adenovirus-CD 154 (Ad-ISF35) in Patients With Chronic Lymphocytic Leukemia/ Small Lymphocytic Lymphoma
Brief Title: Study of Repeat Intranodal Injection of Memgen's Cancer Vaccine, Ad-ISF35, in Subjects With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug supply became unavailable
Sponsor: Januario Castro, M.D. (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Memgen, LLC (Industry)
Responsible Party: Sponsor-Investigator, Januario Castro, M.D., Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD-101357 - prev 080497; CLL-35-202
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-ISF35 (Experimental): Ad-ISF35, intranodal injection, 3.3 x 10^10 ISF35 viral particles, every 2-4 weeks up to six total injections.
  Interventions: Biological: ISF35

INTERVENTIONS:
Biological: ISF35 — Subjects participating in this study will be treated with multiple doses of Ad-ISF35 given via intranodal injection using a fixed dose of 3.3 x 10^10 ISF35 viral particles. Intranodal injections will be administered every 2-4 weeks up to six total injections.

SUMMARY:
This is a Phase II, open label, fixed dose, repeat injection, single institution study. Eligible subjects will receive up to six doses of Ad-ISF35 injected directly into a selected lymph node under ultrasound guidance. The primary goal is to determine and monitor clinical and biological responses in patients treated with repeat intranodal injections of Ad-ISF35.

DETAILED DESCRIPTION:
This is a phase II clinical trial in which study subjects will be treated with multiple doses of Ad-ISF35 given via intranodal injection using a fixed dose of 3.3 x 10^10 ISF35 viral particles. Intranodal injections will be administered every 2-4 weeks up to six total injections.

Because this is the first time that repeat administration of Ad-ISF35 will be performed via intranodal injection, and in order to allow sufficient time to evaluate the safety and toxicity of this procedure, we will treat subjects 1 thru 3 at one month intervals and with inpatient admission for 24 hours observation. After subject three receives their second ISF35 injection we will proceed with enrollment of cohorts of four patients per month at one week intervals until study enrollment has been completed. These subjects will be treated as outpatients and will be observed for 3 hours prior to discharge.

ISF35 has already been used in Phase I clinical trials. The trials demonstrated that ISF35 treatment is well-tolerated and patients did not experience any significant or unexpected adverse events. Patients reported flu-like symptoms from ISF35, which disappeared within one to three days.

ISF35 is an abbreviation for Immune Stimulatory Factor 35, an offspring of technology discovered by Dr. Thomas J. Kipps, MD, PhD, Professor, Department of Medicine and Deputy Director for Research,UCSD Moores Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B-cell CLL/SLL including:

   * Lymphocytosis of monoclonal B-cells co-expressing ≥ one B-cell marker (CD19, CD20, or CD23) AND
   * CD5 in peripheral blood or lymph node AND
   * Bone marrow with ≥ 30% mononuclear cells having the CLL/SLL phenotype.
2. Presence of at least ONE single accessible AND palpable lymph node in the cervical, supraclavicular, axillary, or inguinal regions. The size of the lymph nodes must be larger than 2x2 cm in the horizontal and perpendicular axes.
3. Intermediate or High risk, poor prognosis CLL/SLL
4. Indication for treatment as defined by the NCI Working Group Guidelines:

   * Massive (> 6 cm below the left costal margin) or progressive splenomegaly OR
   * Massive lymph nodes or nodal clusters (> 10 cm in longest diameter) OR *Progressive lymphadenopathy OR
   * Grade 2 or 3 fatigue OR
   * Fever ≥ 100.5 degrees F OR
   * Night sweats for greater than 2 weeks without documented infection OR
   * Presence of weight loss ≥ 10% over the preceding 6 months OR
   * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period OR
   * An anticipated doubling time of less than 6 months.
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
   * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy.
5. Males and females 18 years of age and older
6. Laboratory parameters as specified below:

   * Hematologic: Hemoglobin ≥ 10 g/dL (may be post-transfusion); platelet count ≥ 50x10^3/mm^3
   * Hepatic: Total Bilirubin < 2 x ULN, and ALT and AST < 2 x ULN
   * Renal: Creatinine ≤ 2 x ULN
7. ECOG Performance Status ≤ 2
8. Anticipated survival of at least 3 months
9. For men and women of child-producing potential, use of effective barrier contraceptive methods during the study and for one month following treatment.
10. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
11. Negative test results for current/active infection with HIV-1, HIV-2, HTLV-1, HTLV-2, CMV, hepatitis A, B, C within 30 days of registration. (Antibody, antigen and nucleic acid tests acceptable, depending on institutional standards.).
12. Subjects must give written informed consent to participate in this trial.
13. Subjects must have received treatment for CLL with chemotherapy agents or antibodies OR if subjects are previously untreated they must state in the consent form that they are refusing to be treated with chemotherapy or antibodies.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Treatment with chemotherapy or monoclonal antibody within 28 days prior to entering the study.
3. Treatment with chemotherapy or monoclonal antibody during the time of participation in this trial.
4. Grade 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
5. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, COPD).
6. Participation in any investigational drug study within 28 days prior to ISF35 administration. (Patient must have recovered from all acute effects of previously administered investigational agents)
7. History of malignancy other than CLL within five years of registration, except patients with adequately treated basal, squamous cell carcinoma or localized cervical cancer.
8. Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis.
9. Any illness or condition that in the opinion of the Investigator may affect safety of treatment or evaluation of any the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, M.D., Principal Investigator — Associate Clinical Professor in the Blood and Marrow Transplantation Division; Thomas J Kipps, M.D., Ph.D., Principal Investigator — Professor of Medicine, Evelyn and Edwin Tasch Chair in Cancer Research in the UCSD School of Medicine
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ad-ISF35
Started | 6
Completed | 3
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Determine and Monitor Clinical and Biological Responses in Patients Treated With Repeat Intranodal Injections of Ad-ISF35.
Time Frame: 2 years (evaluation will be approx. 4 months per patient)
Population: The study was not completed due to unavailability of the study drug, and therefore data were not collected for this Outcome Measure.
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine the Safety of Repeat Administration of Ad-ISF35 Injected Directly Into Lymph Nodes of Patients With CLL/SLL.
Time Frame: 2 years (evaluation will be approx. 1 year per patient)
Population: as for outcome 1
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine Pharmacodynamic Parameters in Patients Treated With Repeat Intranodal Injections of Ad-ISF35.
Time Frame: 2 years (evaluation will be approx. 4 months per patient)
Population: as for outcome 1
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ad-ISF35
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ad-ISF35 (N=6)
Hyponatremia (General disorders) | 1
Flu like syndrome (Immune system disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Fever (General disorders) | 6
Arthritis (non-septic) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Injection site reaction (Immune system disorders) | 6
Sweating (General disorders) | 6
Fatigue (General disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Dyspnea-Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2
Anorexia (General disorders) | 3
Urinary frequency (Renal and urinary disorders) | 2
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes